CLINICAL TRIAL: NCT06260761
Title: Clinical Results of Minimally Invasive Plate Osteosynthesis Versus Conventional Approach in Volar Locking Plate for Close Fractures of Distal End Radius Under WALANT
Brief Title: MIPO Versus Conventional Approach in Volar Locking Plate for Close Fractures Distal End Radius Under WALANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Police General Hospital, Thailand (Other)
Responsible Party: Principal Investigator, Suphasan Keatisuwan, Principal Investigator, Police General Hospital, Thailand
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dh3108103/64
Record Dates: First submitted 2024-01-25; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Radius; Fracture, Lower or Distal End
Keywords: MIPO; distal end radius fracture; WALANT
MeSH Terms: conditions — Fractures, Bone | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: prospective, parallel group, assessor-blinded, randomized controlled trial. randomized with computer generator number and use block-of-four.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The data collector, an orthopedic resident unaware of the surgical technique used, obtained information after operation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIPO (Experimental): isolated close fracture of distal end radius
  Interventions: Procedure: MIPO
- Conventional (Active Comparator): isolated close fracture of distal end radius
  Interventions: Procedure: Conventional

INTERVENTIONS:
Procedure: MIPO — minimal invasive surgery with Volar locking plate fixation in isolated close fracture of distal radius under WALANT
  Arms: MIPO
Procedure: Conventional — standard surgery with Volar locking plate fixation in isolated close fracture of distal radius under WALANT
  Arms: Conventional

SUMMARY:
The goal of this clinical trial is to compare the Minimally Invasive Plate Osteosynthesis (MIPO) approach with conventional methods in volar locking plate treatment for distal end radius fractures under the Wide Awake Local Anesthesia No Tourniquet (WALANT) technique. The main question it aims to answer is: Does the MIPO approach provide better pain control than the conventional approach of volar locking plate fixation in distal radius fractures under WALANT? Participants will be requested to record their pain on the Visual Analog Scale (VAS), assess their functional scores, and undergo postoperative radiographic evaluations. Researchers will compare the MIPO group and the conventional group to determine the postoperative pain VAS scores, shedding light on the comparative effectiveness of the two approaches.

DETAILED DESCRIPTION:
Gap of knowledge

* No comparison of conventional Versus MIPO technique under WALANT
* No result in acute post-operative pain

ELIGIBILITY:
Inclusion Criteria:

* isolated closed fractures of the distal end radius requiring surgery
* aged 18 years and older

Exclusion Criteria:

* Patients with bone fractures lasting more than 21 days
* open fractures
* articular multi-fragmentary comminuted fractures of the distal radius
* not suitable to undergo volar approach surgery
* individuals with combined carpal fractures or dislocation
* ulna fractures
* associated injuries
* a history of previous wrist surgery
* diabetes mellitus
* chronic wrist inflammation
* wrist bone deformities
* the use of anticoagulation drugs
* uncooperative behavior
* those refusing to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2023-02-05 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Pain Visual analogue scale | Postoperative day 0-7 and 2,6,10,14,24 weeks
  pain 0-10, minimum = 0 (best) , maximum = 10 (worst)

SECONDARY OUTCOMES:
Quick Disabilities of the Arm, Shoulder and Hand | Postoperative 2,6,10,14,24 weeks
  functional score 0-100 , minimum = 0 (best) , maximum = 100 (worst)
Grip strength | Postoperative 2,6,10,14,24 weeks
  compare with normal side 0-100%
Pinch strength | Postoperative 2,6,10,14,24 weeks
  compare with normal side %
Range of motion | Postoperative 2,6,10,14,24 weeks
  flexion extension pronation supination ulnar and radial deviation (degree)
Aesthetics | Postoperative 24 weeks
  range 0-5; 0=bad 3=so so 5=good
Satisfy | Postoperative 24 weeks
  range 0-5; 0=Unsatisfied 3=so so 5=Satisfy
Volar tile | Postoperative 2, 24 weeks
  radiographic parameter (degree)
ulnar variance | Postoperative 2, 24 weeks
  radiographic parameter (centimeter)
radial inclination | Postoperative 2, 24 weeks
  radiographic parameter (degree)
operation time | Intraoperative
  (minute)
skin incision | Postoperative 2 weeks
  (centimeter)
morphine IV use | Postoperative day 0-2
  (milligram)
complication | up to 24 weeks
  Number of Participants with complication and adverse event

CONTACTS AND LOCATIONS:
Overall Officials: suphasan keatisuwan, M.D., Principal Investigator — Police general hospital, Bangkok, Thailand
Locations (1):
- Police general hospital, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pire E, Hidalgo Diaz JJ, Salazar Botero S, Facca S, Liverneaux PA. Long Volar Plating for Metadiaphyseal Fractures of Distal Radius: Study Comparing Minimally Invasive Plate Osteosynthesis versus Conventional Approach. J Wrist Surg. 2017 Aug;6(3):227-234. doi: 10.1055/s-0037-1599791. Epub 2017 Mar 16. PMID 28725505
- [Result] Vernet P, Gouzou S, Hidalgo Diaz JJ, Facca S, Liverneaux P. Minimally invasive anterior plate osteosynthesis of the distal radius: A 710 case-series. Orthop Traumatol Surg Res. 2020 Dec;106(8):1619-1625. doi: 10.1016/j.otsr.2020.04.024. Epub 2020 Nov 3. PMID 33153957
- [Result] Zenke Y, Sakai A, Oshige T, Moritani S, Fuse Y, Maehara T, Nakamura T. Clinical results of volar locking plate for distal radius fractures: conventional versus minimally invasive plate osteosynthesis. J Orthop Trauma. 2011 Jul;25(7):425-31. doi: 10.1097/BOT.0b013e3182008c83. PMID 21464735
- [Result] Zhang X, Huang X, Shao X, Zhu H, Sun J, Wang X. A comparison of minimally invasive approach vs conventional approach for volar plating of distal radial fractures. Acta Orthop Traumatol Turc. 2017 Mar;51(2):110-117. doi: 10.1016/j.aott.2017.02.013. Epub 2017 Feb 27. PMID 28246046

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT06260761/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT06260761/ICF_001.pdf